CLINICAL TRIAL: NCT04509336
Title: Comparison of the Efficacy and Safety of Orphenadrine Versus Baclofen in Treatment of Muscle Cramps in Cirrhotic Patients
Brief Title: Orphenadrine Versus Baclofen in Treatment of Muscle Cramps in Cirrhotic Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID 19 Pandemic
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Noha Mansour, Lecturer of clinical pharmacy, pharmacy practice department, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-87
Record Dates: First submitted 2020-07-21; First posted 2020-08-12 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Orphenadrine; Baclofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- orphenadrine group (Experimental): orphenadrine
  Interventions: Drug: Orphenadrine
- Baclofen group (Active Comparator): Baclofen
  Interventions: Drug: Baclofen

INTERVENTIONS:
Drug: Orphenadrine — 100 mg twice daily
  Arms: orphenadrine group
Drug: Baclofen — initial dose of 10 mg tablet once daily, dose will be gradually increased according to the patients responses
  Arms: Baclofen group

SUMMARY:
Muscle cramps are commonly affects patients with cirrhosis. It adversely influences the quality of life of cirrhotic patients. Treatment of muscle cramps still challenging owing to the diversity of the responsible pathophysiological mechanisms.The effectiveness of baclofen and orphenadrine in controlling muscle cramps in cirrhotic patients has been presented in recent randomised controlled clinical trials;however, the comparative efficacy and safety between these two therapeutic options has not been previously investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years
2. Cirrhotic patients complaining of frequent muscle cramps (>3 per week) for at least a month

Exclusion Criteria:

1. Patients with allergy to study drugs
2. Renal impairment
3. Peripheral vascular disease
4. Peripheral neuropathy
5. Glaucoma
6. Prostatic enlargement
7. Pregnancy and lactation
8. Patients taking calcium channel blockers, and conjugated estrogens
9. Patients taking vitamin E, taurine, carnitine, narcotic pain medications, muscle relaxants, nonsteroidal anti-inflammatory drugs, or antispastic agents during and for 2 weeks following the study
10. Patients with alcoholic cirrhosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
the difference in the number of muscle cramps between the orphenadrine and baclofen groups at the end of treatment | 12 weeks
  Questionnaire

SECONDARY OUTCOMES:
The difference in severity of cramps between orphenadrine and baclofen groups at the end of treatment | 12 weeks
  Visual analogue scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Assem Elfert, Study Chair — Tanta University; Sherif Abd-Elsalam, Principal Investigator — Tanta University
Locations (1):
- Tanta University Hospitals, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No